CLINICAL TRIAL: NCT06317467
Title: Characterization of the Physiological and the Pathological Role of Anti-C1q Autoantibodies in Pregnancy: a Potential Treatment for Pre-eclampsia to Prevent Fetal Intrauterine Growth Restriction?
Brief Title: Role of Anti-C1q Autoantibodies in Pregnancy
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 01/2023
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Pre-Eclampsia
Keywords: Anti-C1q autoantibodies; Intra Uterine Growth Restriction (IUGR); Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women with physiological pregnancies: Control group
  Interventions: Other: Blood sampling
- Patients diagnosed for PE: hypertension arisen suddenly after the 20th week of pregnancy with associated proteinuria, greater than or equal to 300 mg/24 hours often corresponding to 30 mg/dL (1+) on a single sample
  Interventions: Other: Blood sampling
- Women affected by SLE, APS, or autoimmune thyroiditis: Patients attending the medically assisted procreation department or the Department of Rheumatology, Division of Internal Medicine, University Medical Centre Ljubljana, Ljubljana, Slovenia
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Four blood samples will be collected, in conjunction with the collection of samples already programmed for assistance during pregnancy: blood sampling for the B-test (within the 13th week of gestation), at the blood test centre of the Institute for Maternal and Child Health, IRCCS Burlo Garofolo; blood sampling for toxoplasmosis or blood sugar level, upon execution of the morphological ultrasound scanning (around the 20th and 34th weeks of gestation), at the blood test centre of the Institute for Maternal and Child Health, IRCCS Burlo Garofolo, as well. Finally, 40 days after delivery, during routine gynaecological control after the puerperium.
Other: Blood sampling — For patient of group 2, the blood sample will be collected at the time of the diagnosis of PE and 40-50 days after delivery in Obstetrics and Gynaecology Department of the institute or in Department of Biomedical Sciences, IRCCS Humanitas Research Hospital, Rozzano, Milan, Italy.

SUMMARY:
Preeclampsia (PE) is a very frequent obstetric complication. C1q, the first recognition molecule of the classical pathway of complement system (C), represents a double-edged molecule in determining pregnancy outcomes. In animal models, C1q deficiency caused the development of a dysfunctional placenta and PE-like symptoms. Conversely, lower levels of C components were detected in the sera of patients with PE due to C consumption and increased deposition of activated C components in the placenta, as well as to the binding to placental apoptotic bodies, syncytiotrophoblast microvesicles (STBM) and debris which are increased in the circulation of patients with PE.

C1q is a hexameric glycoprotein of 460kDa composed by six copies of three polypeptide chains A, B and C, each made by a C-terminal globular head (gC1q) and a N-terminal collagen-like region (CLR). This molecule can be the target of an antibody response. Autoantibodies targeting C1q were first recognized in the serum of Systemic Lupus Erythematosus (SLE) patients. The presence of anti-C1q autoantibodies was also detected in patient affected by autoimmune disease (ie, kidney disorders, vasculitis, thyroiditis). Almost all of these autoimmune disorders are associated with an increased risk of developing PE during pregnancy.

Anti-C1q detection mainly concerns the prediction of the onset of lupus nephritis (LN) in SLE patients. Although anti-C1q autoantibodies do not deplete circulating C1q, their presence in maternal circulation and in placenta may trigger improper C activation and impair C1q activity. In pregnancies complicated by autoimmune affection such as SLE, autoimmune thyroid disorders and Antiphospholipid syndrome (APS) the prevalence of anti-C1q appeared to be higher than in control pregnancies and associated with miscarriage. High levels of anti-C1q have been found in a group of Japanese patients suffering recurrent pregnancy loss (RPL). In a group of anti-C1q positive healthy pregnancies and LN patients was assessed whether C1q autoantigenic behaviour could vary among individuals with or without correlated manifestation. Sera from healthy pregnancies and LN patients were screened for the presence of autoantibodies against the CLR fragment and/or the gC1q: antibodies against gC1q were found in both groups, whereas anti-CLR were only detected in the LN one, suggesting that only the latter may have a pathogenic role. Despite this, the biological functions of anti-C1q remain far from clear

ELIGIBILITY:
Inclusion Criteria Group 1. Women occurring physiological pregnancies that sign the consent to participate in the study and agree to spontaneously return to the maternal hospital 40 days after delivery.

Group 2. Patients diagnosed for PE (hypertension arisen suddenly after the 20th week of pregnancy with associated proteinuria, greater than or equal to 300 mg/24 hours often corresponding to 30 mg/dL (1+) on a single sample).

Group 3. Women affected by SLE, APS, or autoimmune thyroiditis attending the medically assisted procreation department or the Department of Rheumatology, Division of Internal Medicine, University Medical Centre Ljubljana, Ljubljana, Slovenia

Exclusion criteria

1. Women aged under 18 years
2. Viral or bacterial blood transmitted infections.
3. Patients whose informed consent cannot be obtained.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women, women attending the medically assisted procreation
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Between groups difference in percentage of anti-gC1q compared to the total anti-C1q autoantibodies | 8-12 weeks of gestation
Between groups difference in percentage of anti-cC1q compared to the total anti-C1q autoantibodies | 8-12 weeks of gestation
Between groups difference in percentage of anti-gC1q compared to the total anti-C1q autoantibodies | 20-24 weeks of gestation.
Between groups difference in percentage of anti-cC1q compared to the total anti-C1q autoantibodies | 20-24 weeks of gestation.
Between groups difference in percentage of anti-gC1q compared to the total anti-C1q autoantibodies | 34-38 weeks of gestation.
Between groups difference in percentage of anti-cC1q compared to the total anti-C1q autoantibodies | 34-38 weeks of gestation.
Between groups difference in percentage of anti-gC1q compared to the total anti-C1q autoantibodies | 40-50 days after delivery.
Between groups difference in percentage of anti-cC1q compared to the total anti-C1q autoantibodies | 40-50 days after delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided